CLINICAL TRIAL: NCT04784169
Title: Free Middle Turbinate Flap for Repair of Low Flow Cerebrospinal Fluid Leak
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Qiangping Wang, MD, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20210086
Record Dates: First submitted 2021-01-08; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: CSF Leakage
MeSH Terms: conditions — Cerebrospinal Fluid Rhinorrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- free middle turbinate flap group (Experimental): A free middle turbinate flap is used to repair the leakage
  Interventions: Device: free middle turbinate flap
- vascularized nasoseptal flap (Active Comparator): A vascularized nasoseptal flap is used to repair the leakage
  Interventions: Device: vascularized nasoseptal flap

INTERVENTIONS:
Device: free middle turbinate flap — Repairing low flow leak using free middle turbinate flap
  Arms: free middle turbinate flap group
Device: vascularized nasoseptal flap — Repairing low flow leak using fascia lata
  Arms: vascularized nasoseptal flap

SUMMARY:
Limited literature has been reported the use of free middle turbinate flap during an endoscopic approach to treat cerebrospinal fluid (CSF) leak, and the results were inconclusive. The overall purpose of this study was to assess the efficacy and safety of free middle turbinate flap in reparing CSF leak during an endoscopic approach.

DETAILED DESCRIPTION:
Cerebrospinal fluid (CSF) rhinorrhea results from an abnormal communication between the sinonasal cavity and the subarachnoid space. It may occur spontaneously or secondary to accidental or iatrogenic trauma. CSF leak is a potentially devastating condition that can lead to ascending meningitis, pneumocephalus, and intracranial abscess. Surgical repair is recommended for most patients with CSF leaks to prevent the potential sequelae.

Multiple graft materials have been employed in the approach, including temporalis fascia, middle turbinate flap, fascia lata, fat, free cartilage or bone, vascularized nasoseptal flap and acellular skin grafts. Among these options, vascular nasoseptal ﬂaps are the most popular materials at present. Limited literature has been reported the use of free middle turbinate flap during an endoscopic approach to treat CSF rhinorrhea, and the results were inconclusive. There were a large number of cases using free middle turbinate flap for CSF rhinorrhea repair in our institution. The purpose of this study was to determine the efficacy and safety of the free middle turbinate flap for repair of CSF rhinorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing repairing of CSF leak under transsphenoidal approach
* Dural defect smaller than 1cm
* No extensive arachnoid dissection
* No dissection into a ventricle or cistern

Exclusion Criteria:

* High flow CSF leak

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Cerebrospinal Fluid (CSF) Leak | 1month

SECONDARY OUTCOMES:
Number of Participants With Postoperative Complications | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GAO HUI, Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- GAO HUI, Wuhan, Hubei, China